CLINICAL TRIAL: NCT06890247
Title: Single-dose Intra-Articular of a Hybrid Purified Hyaluronic Acid with a High Molecular Weight and Sodium Chondroitin of Biotechnological Origin in Combination with Rehabilitation Treatment in Sports Adults with Osteoarthritis of the Knee
Brief Title: Single-Dose Hybrid Hyaluronic Acid and Sodium Chondroitin with Rehabilitation for Sports Adults with Knee Osteoarthritis
Status: Not yet recruiting | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof.ssa Giulia Letizia Mauro, Professor, University of Palermo
Other Study IDs: MFR042025
Record Dates: First submitted 2025-03-16; First posted 2025-03-21 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; Knee; Hyaluronic Acid; Sodium Chondroitin; Rehabilitation; Sports Adults; Isokinetic Testing; Pain Relief; Functional Improvement
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
: This observational case-control study aims to evaluate the efficacy of a single-dose intra-articular injection of a hybrid purified hyaluronic acid with high molecular weight and sodium chondroitin of biotechnological origin, combined with rehabilitation treatment, in sports adults with moderate to severe knee osteoarthritis. Additionally, the study incorporates isokinetic testing to assess muscle strength and functional capacity.

The primary objective is to determine whether this combined treatment improves pain relief, functional capacity, and overall quality of life compared to rehabilitation treatment alone. Participants aged 18 to 50 years, diagnosed with knee osteoarthritis, will be recruited from clinics at the U.O.C. of Recovery and Functional Rehabilitation at A.O.U.P. P. Giaccone in Palermo. Participants will be divided into two groups: one receiving the hybrid hyaluronic acid and sodium chondroitin injection along with rehabilitation, and the other receiving only rehabilitation. The study will also utilize isokinetic testing to provide objective measurements of muscle strength and endurance.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 50 years.
* Radiologically confirmed diagnosis of knee osteoarthritis (Kellgren-Lawrence grade ≤3), present for at least 6 months.
* Persistent moderate to severe pain due to osteoarthritis, interfering with physical performance.
* Documented reduction in sports performance (use appropriate scales or tests to validate this).
* Lack of response to pharmacological or other conservative treatments.
* Willingness to provide written informed consent for participation.

Exclusion Criteria:

* Coexisting rheumatic diseases.
* History of intra-articular viscosupplementation in the target knee within the previous 6 months.
* Presence of significant venous or lymphatic stasis.
* Body Mass Index (BMI) ≥ 30 kg/m².
* Use of systemic or intra-articular corticosteroids in the target knee within the last 3 months.
* Chronic use of topical/systemic analgesics, NSAIDs, or narcotics.
* History of alcohol or drug abuse.
* Allergy or hypersensitivity to hyaluronic acid or any of its components.
* Pregnant or breastfeeding women, or those not using adequate contraception.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants will be recruited from the outpatient clinics of the Unit of Recovery and Functional Rehabilitation at the A.O.U.P. P. Giaccone Hospital in Palermo. The study focuses on sports-active adults aged 18 to 50 years with clinically and radiologically confirmed knee osteoarthritis, seeking treatment for moderate to severe pain affecting physical performance.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Pain Levels Assessed by the Numerical Rating Scale (NRS) at 90 Days | From baseline (T0) to 90 days (T3) post-intervention
  The primary outcome will assess the change in pain intensity using the Numerical Rating Scale (NRS). This scale ranges from 0 to 10, where 0 indicates no pain and 10 represents the worst possible pain. Pain intensity will be measured at baseline (T0) and at 90 days (T3) following the intervention. The change in NRS scores between these time points will quantify the treatment's effectiveness in reducing knee pain among study participants. Participants with a clinically meaningful reduction in pain (defined as a decrease of at least 2 points on the NRS) will be considered responders.

SECONDARY OUTCOMES:
Change from Baseline in Functional Capacity Assessed by Lequesne Index at 30 and 90 Days | Baseline (T0), 30 days (T2), and 90 days (T3).
  Evaluation of changes in the Lequesne Index, a validated tool that measures functional disability in knee osteoarthritis patients. The index assesses pain, maximum walking distance, and daily activities. Scores range from 0 (no disability) to a maximum score indicating severe disability. Higher scores denote worse functional impairment. Measurements will be recorded at baseline (T0), 30 days (T2), and 90 days (T3).
Change from Baseline in Quality of Life Assessed by SF-12 Questionnaire | Baseline (T0) and 90 days (T3).
  Assessment of changes in quality of life using the SF-12 Health Survey, which evaluates both physical and mental health components. The SF-12 generates composite scores for these domains, with higher scores indicating better quality of life. Measurements will be taken at Baseline (T0) and compared to 90 days (T3) post-intervention to assess the impact of the treatment.
Change from Baseline in Muscle Strength Evaluated with Isokinetic Testing | Baseline (T0) and 90 days (T3).
  Measurement of muscle strength parameters, including peak torque, endurance, and total work of the knee flexor and extensor muscles, using isokinetic dynamometry. Testing will be performed at three angular velocities (0°, 60°, and 120°/sec). Data collected at Baseline (T0) will be compared to follow-up measurements at 90 days (T3) to evaluate the functional improvement in muscle performance.

CONTACTS AND LOCATIONS:
Locations (1):
- A.O.U.P. P. Giaccone, Palermo, Italia, Palermo, Italia, Italy